

## Ministry Of Health Nineveh Health Directorate Training & Human Development Center



Decision number: (79/21)

Date: 2021/7/11

Form number 2021/03

ch committee decision

The research committee of Nineveh Health Directorate has discussed the research protocol number (79/21)

## Entitled:

(Assessment of three years follow up to rehabilitative program for patients with Spinal Cord Injury from Sab-acute stage to Ambulation).

Submitted by researchers:

(Munib Abdullah Fathe, Wassim Moalla, Saad Kazim Karim)

To the research and knowledge management unit at the training and human development center of Nineveh Health Directorate on Mosul /Iraq

## The committee has decided to:

\*Accept the above-mentioned research protocol as it meets the standards adopted by ministry of health for the implementation of research, and there is no objection to implementing it in the directorate's institution.

Rapporteur of the committe

Dr. Marab Younis Abdullh Al-Pat

Chairman of the committee Dr. Muataz Abdul-Aljawad Al-Aani

## Notes:

- The committee chairperson / committee rapporteur was authorized to sign this decision on behalf of the remaining members of the committee under the rules of procedure of the research committee.
- -The Research Committee approval means that the research project submitted to the aforementioned committee has fulfilled the ethical and methodological standards adopted by the Ministry of Health for conducting a research. As for the Implementation of the research, it depends on the researcher's adherence to the Instructions of the health institution in which the research will be implemented as well as the laws, instructions and recommendations in force that govern the practice of medical and health action in Iraq.